CLINICAL TRIAL: NCT01088698
Title: Prospective Study of the Combination of Golimumab and UVB-311nm Phototherapy in Patients With Psoriatic Arthritis and Psoriatic Skin Lesions
Brief Title: Golimumab Plus UVB-311nm in Psoriasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruiting patients;
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Peter Wolf, MD, Professor of Bioimmunotherapy, Medical University of Graz
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-110 ex 09/10
Record Dates: First submitted 2010-03-15; First posted 2010-03-17 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Psoriasis
Keywords: psoriasis; golimumab; TNF-alpha inhibition; phototherapy; 311-nm
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: UVB-311nm radiation — UVB-311nm radiation given 3 times a week to one randomized body-half
  Other Names: narrow-band UVB radiation

SUMMARY:
Golimumab, a TNF-alpha antibody, has been approved in the EC and USA for the treatment of psoriatic arthritis. The aim of this study is to determine in a randomized half-side comparison whether additional narrowband UVB-311nm phototherapy accelerates and improves the clearance of psoriatic skin lesions in golimumab-treated patients.

DETAILED DESCRIPTION:
Psoriatic skin lesions of patients with psoriatic arthritis who receive standard treatment with golimumab (50 mg or 100 mg s.c. once a month depending on total body weight whether below or above 100 kg, respectively) are exposed to UVB-311nm phototherapy on a randomized body half (left or right; head exempt) 3 x per week for six weeks and/or until complete response (defined as reduction in PASI to < 3). A patient qualifies if A) golimumab was started within a week or B) after 3 months of golimumab treatment the PASI reduction is smaller than 90%. PASI score, patient visual analogue score (VAS) for therapeutic response, and patient VAS for severity of skin lesions is assessed weekly; and at follow-up visits at month 3, 6, and 12. The primary hypothesis is that phototherapy increases the PASI reduction on the exposed body site by more than 20%. Paired Wilcoxon testing for differences in PASI and patient VAS scores is done; Fisher exact test is applied to determine differences in complete remission, PASI reduction > 90%, > 75% and/or 50% between body sites.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients with psoriatic arthritis who receive treatment with golimumab
* Patient wish for treatment of psoriatic skin lesions

Exclusion Criteria:

* Pregnancy or lactation
* Presence and/or history of malignant melanoma
* Presence and/or history of invasive squamous cell carcinoma of the skin
* Presence and/or history of more than 3 basal cell carcinomas
* Dysplastic nevus syndrome
* Antinuclear antibodies (ds-DNA, Ro/SSA, La/SSB)
* Autoimmune disorders such as lupus erythematosus or dermatomyositis
* Abnormal photosensitivity and photosensitive diseases such as porphyria, chronic actinic dermatitis, Xeroderma pigmentosum, basal cell nevus syndrome, and others
* General poor health status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Psoriasis area and severity index (PASI) reduction from baseline comparing the UV-irradiated vs. the non-irradiated body site | week 6
  The effect of treatment on PASI will be determined. The primary hypothesis is that UVB-311nm treatment leads to a difference in the reduction of PASI from baseline by > 20% comparing the UV-irradiated vs. the non-irradiated body site at week 6 of treatment.

SECONDARY OUTCOMES:
Patient visual analogue (VAS) score for the therapeutic effect and severity of skin lesions | week 6

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Medical University of Graz, Austria
Locations (1):
- Medical University of Graz, Graz, Austria